CLINICAL TRIAL: NCT07240142
Title: Biochemical and Docking Evidence of Neurotransmitter Dysregulation in Specific Learning Disorder
Brief Title: Neurotransmitter Levels in Children With Specific Learning Disorder
Acronym: SLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilara Ulger Ozbek (Other)
Responsible Party: Sponsor-Investigator, Dilara Ulger Ozbek, Dr., Cumhuriyet University
Organization: Cumhuriyet University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCÜ Child Psychiatry
Record Dates: First submitted 2025-09-30; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Specific Learning Disability; Healthy (Controls)
Keywords: Specific learning Disorder; Glutamate; L-arginine; nitric oxide; molecualr docking
MeSH Terms: conditions — Specific Learning Disorder

STUDY DESIGN:
Intervention Model Description: Blood sample collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of blood samples (Experimental): A 5 ml blood sample will be taken from the left arterial vein of the individuals in the study group, and serum will be obtained from it. The neurotransmitter concentrations specified in the serum samples will be measured with an ELISA test kit.
  Interventions: Procedure: Blood Product; Other: Elisa test

INTERVENTIONS:
Procedure: Blood Product — Collecting 5 ml blood samples from the left atrial vein, after that obtaining serum from it.
Other: Elisa test — Measurement of glutamate, nitric oxide, and L-arginine concentrations in the blood samples obtained using an ELISA test kit.

SUMMARY:
The aim of this clinical trial was to measure how specific neurotransmitter levels in children with Specific Learning Disorder (SLD) change compared to controls. The relationship between these markers and the measured markers will be determined both theoretically and experimentally using various neuropsychological tests. The fundamental questions it aims to answer are

Did neurotransmitter levels increase or decrease in the patient group? Are the neurotransmitter levels measured in the neuropsychological tests related? Can the measured neurotransmitters be used to predict the disease?

Participants:

A single visit to the clinic, a blood sample, and neuropsychological tests will be administered on the same day.

DETAILED DESCRIPTION:
The purpose of this investigation was to assess the levels in serum of key neurotransmitters and their precursors (glutamate, L-arginine, and nitric oxide) in children with SLD and also to integrate these biochemical results with molecular docking analyses of their interactions with phospholipase A2 (PLA2) and N-methyl D-aspartate receptors (NMDA), both of which play significant roles in learning function in these patients.

The research group consisted of 20 children aged 7-14 years who had been diagnosed with SLD using DSM-5 criteria, as well as 20 age-matched, gender-matched, and educationally matched healthy controls. The children in the study group underwent the Stroop Test [Total Error Scores, Total Time Scores, Total Correction] and the Wechsler Intelligence Scale for Children (WISC-IV) subtests, and the results were scored. The serum concentrations of glutamate, L-arginine, and nitric oxide (NO) were determined using ELISA. The diagnostic ability of the biomarkers was evaluated using ROC analysis. Additionally, the interactions of glutamate and L-arginine with the PLA2 enzyme and the NMDA receptor were examined using molecular docking analysis.

ELIGIBILITY:
Inclusion Criteria:

* Study group: no additional mental disorder except a specific learning disability,
* The control group had no mental illness.
* Having no head injury or neurological illness for all groups.
* There is no drug that might possibly alter cognitive functions for all populations.

Exclusion Criteria:

* The study group had a mental disease other than a specific learning disability and ADHD.
* The control group had any mental condition.
* Having a head injury or neurological illness in all categories.
* Using drugs that may impair cognitive functioning in all groups those with additional diseases

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Mesurment of serum neurotransmitters levels | 6 months
  Serum Glutamate Levels (measured in µmol/L by ELISA at baseline)
  Serum L-Arginine Levels (measured in µmol/L by ELISA at baseline)
  Serum Nitric Oxide (NO) Levels (measured in µmol/L by ELISA at baseline)
Verbal Comprehension Index (VCI) | 6 month
  Change in Verbal Comprehension Index (VCI) score from baseline to 6 months.Points on a scale (range: 40-160; higher scores indicate better performance)
Perceptual Reasoning Index (PRI) | 6 months
  Change in Perceptual Reasoning Index (PRI) score from baseline to 6 months. Change in Perceptual Reasoning Index (PRI) score from baseline to 6 months.
Working Memory Index (WMI) | 6 months
  Change in Working Memory Index (WMI) score from baseline to 6 months. Points on a scale (range: 40-160; higher scores indicate better performance)
Processing Speed Index (PSI) | 6 months
  Change in Processing Speed Index (PSI) score from baseline to 6 months. Points on a scale (range: 40-160; higher scores indicate better performance).
Stroop Test Performance | 6 months
  Change in Stroop Test total errors, total time, and total corrections from baseline to 6 months.Seconds (for time) and number of errors/corrections; lower scores indicate better performance.
Full Scale IQ (FSIQ) | 6 months
  Change in Full Scale IQ (FSIQ) score from baseline to 6 months.oints on a scale (range: 40-160; higher scores indicate better performance)

OTHER OUTCOMES:
Molecular docking analysis | 6 months
  Binding affinity values (in kcal/mol) of Glutamate and L-Arginine ligands to NMDA receptor and PLA2 enzyme active sites will be evaluated using molecular docking analysis. Lower binding affinity (more negative kcal/mol) indicates stronger interaction.Lower (more negative) binding energy indicates a stronger binding affinity.
ROC analysis performance of biomarkers | 6 months
  Receiver Operating Characteristic (ROC) analysis will be performed to determine the diagnostic performance of selected biomarkers. Parameters include Area Under the Curve (AUC), sensitivity, specificity, cut-off value, and Youden Index. AUC value (range 0-1); higher values indicate better diagnostic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara ULGER OZBEK, Dr., Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No